CLINICAL TRIAL: NCT04301817
Title: Changes in Optic Nerve Sheath Diameter in Patients Undergoing Spinal Surgery in the Prone Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 20200305
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Optic Nerve Sheath Diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prone position: Patients undergoing surgery in prone position

SUMMARY:
Long standing prone position could affect vision or optic nerve. To measure the optic nerve sheath diameter using ultrasound is quick and useful assessments of patients.

This study will look at the change of optic nerve sheath diameters of patients undergoing surgery in prone position

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery in prone position

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients has ophthalmic diseases
* Patients has previous history of ophthalmic surgery.
* Patients has neurological disorders.
* Patients has history of head surgery.
* Severe anaphylactic allergy to ultrasound gel or Tegaderm

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing prone position surgery in out institute.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change optic nerve sheath diameter | 0,1,3,6,24 and 48 hours
  Change in Optic nerve sheathe diameter from baseline, before surgery, immediate after surgery (prone, supine), 1,3,6,24 and 48 hours after completion of surgery

REFERENCES:
- [Result] Yu J, Hong JH, Park JY, Hwang JH, Cho SS, Kim YK. Propofol attenuates the increase of sonographic optic nerve sheath diameter during robot-assisted laparoscopic prostatectomy: a randomized clinical trial. BMC Anesthesiol. 2018 Jun 20;18(1):72. doi: 10.1186/s12871-018-0523-7. PMID 29925316
- [Result] Chin JH, Seo H, Lee EH, Lee J, Hong JH, Hwang JH, Kim YK. Sonographic optic nerve sheath diameter as a surrogate measure for intracranial pressure in anesthetized patients in the Trendelenburg position. BMC Anesthesiol. 2015 Mar 31;15:43. doi: 10.1186/s12871-015-0025-9. eCollection 2015. PMID 25861241